CLINICAL TRIAL: NCT07039019
Title: Pilot, RandOmized Study of the Feasibility and Efficacy of PrednisonE for Non-specifiC pleuriTis
Brief Title: Study of the Feasibility and Efficacy of PrednisonE for Non-specifiC pleuriTis
Acronym: PROSPECT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Udit Chaddha, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY-25-00427
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Pleuritis, Non-specific
MeSH Terms: conditions — Pleurisy | interventions — Adrenal Cortex Hormones; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with Corticosteroids (Experimental): Standard of care (corticosteroids) as per institutional practice. If the treatment is effective, patients continue for another 4 weeks while taking medication to prevent infections. If it's not effective, they begin a gradual dose reduction until stopping.
  Interventions: Drug: Corticosteroid
- Patients with No Corticosteroids (Active Comparator): Patients will not receive any corticosteroids.
  Interventions: Other: No Corticosteroid

INTERVENTIONS:
Drug: Corticosteroid — Patients take 40 mg of prednisone daily for 4 weeks to help reduce inflammation.
  Other Names: Prednisone
  Arms: Patients with Corticosteroids
Other: No Corticosteroid — Patients do not take corticosteroid.
  Arms: Patients with No Corticosteroids

SUMMARY:
This research study aims to evaluate whether corticosteroids help prevent the recurrence of pleural effusions in patients with non-specific pleuritis diagnosed through pleural biopsy. It can lead to recurrent fluid buildup in the lungs, causing discomfort and requiring additional medical interventions. There is no established treatment to prevent recurrence, and this study seeks to determine whether steroids reduce fluid buildup or cause complications.

There will be two groups: one receiving corticosteroids (standard of care in the institution) and one not receiving corticosteroids (intervention group). The participation will last approximately 6 months, with in-person visits every 2 weeks for the first month, then monthly, along with possible telephone follow-ups. The study will monitor for pleural effusion recurrence, need for additional procedures, and potential side effects of corticosteroids.

This is a pilot study. Although there are forty people expected to take part in this research study based on institutional data, the number of patients included in the study will be determined by the number of patients with non-specific pleuritis diagnosed during the study period.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with diagnosis of non-specific pleuritis as determined by pleural biopsy with a negative serologic autoimmune profile (ANA, ANCA, anti-DS DNA, anti-SS A/B, anti-centromere, RF, anti-CCP) are eligible

Exclusion Criteria:

* Chronic/fibrinous pleuritis
* Positive autoimmune serologic workup
* A contraindication to corticosteroids
* Empyema
* Patients already receiving corticosteroids or other immunosuppressive medications for any other indication
* Inability to obtain informed consent due to cognitive, neurologic or psychiatric impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-11-19 (Estimated); Study Completion 2026-11-19 (Estimated)

PRIMARY OUTCOMES:
Number of patients screened | every 2 weeks after pleuroscopy for the first 4 weeks, and then monthly up to 6 months
  Screened defined as how many patients are evaluated for participation
Number of patients enrolled | every 2 weeks after pleuroscopy for the first 4 weeks, and then monthly up to 6 months
  Enrolled defined as how many screened patients actually join the study
Number of patients retained | every 2 weeks after pleuroscopy for the first 4 weeks, and then monthly up to 6 months
  Retention defined as how many enrolled patients continue participating over time

SECONDARY OUTCOMES:
Rate of recurrence | every 2 weeks after pleuroscopy for the first 4 weeks, and then monthly up to 6 months
  Incidence of recurrent pleural effusions attributable to symptoms requiring an intervention

CONTACTS AND LOCATIONS:
Overall Officials: Udit Chaddha, MBBS, Principal Investigator — Icahn School of Medicine
Locations (2):
- United States (2):
  - Mount Sinai Hospital, New York, New York
  - Mount Sinai Morningside, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Proposals should be directed to udit.chaddha@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (link to be determined).